CLINICAL TRIAL: NCT00726284
Title: BIOMET/EBI (Electro-Biology, Inc) Spine Patient Outcomes Registry
Brief Title: Spine Patient Outcomes Registry for Biomet/EBI (Electro-Biology, Inc)
Acronym: SPO
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-006
Record Dates: First submitted 2008-07-29; First posted 2008-07-31 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Degenerative Disc Disease; Spinal Stenosis
Keywords: Herniated nucleus pulposus (HNP)
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this patient registry is to prospectively collect data on patients who are having spinal surgery with EBI and Interpore Cross Spine Products.

DETAILED DESCRIPTION:
A patient registry to prospectively collect data on patients who are having spinal surgery with EBI and Interpore Cross Spine Products.

ELIGIBILITY:
Inclusion Criteria:

N/A

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This is an open cohort prospective patient registry conducted at multiple clinical centers
Sampling Method: Non-Probability Sample
Enrollment: 651 (Actual)
Dates: Start 2004-04; Primary Completion 2007-12-06 (Actual); Study Completion 2007-12-06 (Actual)

PRIMARY OUTCOMES:
Fusion Status | 24 Months
  The primary outcome measure for this trial will be the percentage of successful fusions achieved.

SECONDARY OUTCOMES:
Mean VAS (Visual Analog Scale) Score Change from baseline | 24 Month
Oswestry Disability Index / Neck Disability Index (which ever is appropriate for the subject) change from baseline | 24 Month
neurologic Assessment - maintenance or Improvement | 24 Month
SF-36 (Short Form Survey-36) Health Outcomes - Change from Baseline | 24 Month

CONTACTS AND LOCATIONS:
Overall Officials: John Evangelsita, MD, Study Director — EBI, LLC dba Biomet Spine, Biomet Trauma, Biomet Osteobiologics and Biomet Bracing
Locations (5):
- United States (5):
  - Neurological Surgery Associates, Little Rock, Arkansas
  - Florida Orthopedics Association, Orange City, Florida
  - CNS Healthcare, Akron, Ohio
  - Oklahoma Spine and Brain, Tulsa, Oklahoma
  - Pottstown Memorial Medical Center, Pottstown, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided